CLINICAL TRIAL: NCT02316210
Title: Optimization of Onpulse Technology for Patients With Post Surgical or Vascular Oedema
Acronym: TURBO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FKD-TURB-001
Record Dates: First submitted 2014-06-05; First posted 2014-12-12 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Oedema; Neuropathy
MeSH Terms: conditions — Edema | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Digitimer stimulation (Experimental)
  Interventions: Device: electrical stimulation

INTERVENTIONS:
Device: electrical stimulation
  Other Names: Digitimer

SUMMARY:
This study aims to facilitate further optimization of a neuromuscular electrical stimulation device for use in patients whom are suffering from oedema and neuropathy

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and over
2. Be a non-responder to the geko MK1&2 device
3. Able to understand the Subject Information Sheet and willing to sign the written Informed Consent Form.
4. Able and willing to follow the protocol requirements.

Exclusion Criteria:

1. Has a pacemaker
2. Pregnancy.
3. Is contraindicated for the MK1&2 device and/or the Digitimer DS7A
4. Recently diagnosed or suspected DVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Observable foot twitch in response to stimulation with Digitimer DS7A | up to 2 hours
  Upon application of the electrical stimulation, parameters required to achieve an outward deflection of the foot will be measured

SECONDARY OUTCOMES:
adverse events | up to 2 hours
  Any adverse events recorded during the study will be recorded
oedema | up to 2 hours
  oedema will be measured to classify the level of swelling in the participants leg
patient rated tolerability questionnaire | up to 2 hours
  Upon sufficient electrical stimulation to gain an outward deflection of the foot the patient will be asked to complete a tolerability questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- BMI Harbour hospital, Poole, Dorset, United Kingdom